CLINICAL TRIAL: NCT05260229
Title: The Observation About the Effects of Internal Carotid Artery Stenosis on Fundus Vessels and the Changes of Fundus Vessels After Interventional Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: cuiyanqiluteam
Record Dates: First submitted 2022-02-14; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-10

CONDITIONS: Internal Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to collect 30 participants with internal carotid artery stenosis to observed the relationship between the degree of internal carotid artery stenosis and fundus vessels （and blood flow）density before operation, and compared with participants without internal carotid artery stenosis.The fundus blood flow density will be observed after intervention operation in order to see whether the operation is effective to improve the density of fundus vessels and blood flow or not.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with carotid artery stenosis and need surgery;
2. Patients whose vision won't get worse soon;
3. Patients have not had any eye surgeries;
4. Patients with complete profile.

Exclusion Criteria:

1. Patients with severe systemic disease;
2. Patients with poor dioptric stroma;
3. Patients with nystagmus;
4. Patients with incomplete profile.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with carotid artery stenosis and need surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The differences of perfusion density in the Forum of the optical coherence tomography angiography（OCTA ）of Zeiss Company | 2022-01-31
  The perfusion density differences between the fundus vessels（both the macula area and the optic disc area） on the carotid artery stenosis side and the not-significant narrowing side，or the perfusion density differences between the fundus vessels（both the macula area and the optic disc area） on the carotid artery stenosis side and the side with carotid artery stenosis of different degrees.
The differences of perfusion density in the Forum of the optical coherence tomography angiography（OCTA ）of Zeiss Company | 2022-02-14
  The perfusion density differences between the fundus vessels on the carotid artery stenosis side and the same side after interventional surgery.
The differences of vessel density in the Forum of the optical coherence tomography angiography（OCTA ）of Zeiss Company | 2022-01-31
  The vessel density differences between the fundus vessels（both the macula area and the optic disc area） on the carotid artery stenosis side and the not-significant narrowing side，or the vessel density differences between the fundus vessels（both the macula area and the optic disc area） on the carotid artery stenosis side and the side with carotid artery stenosis of different degrees.
The differences of vessel density in the Forum of the optical coherence tomography angiography（OCTA ）of Zeiss Company | 2022-02-14
  The vessel density differences between the fundus vessels on the carotid artery stenosis side and the same side after interventional surgery.
The perimeter and area of the fovea avascular zone（FAZ）in the Forum of the optical coherence tomography angiography（OCTA ）of Zeiss Company | 2022-02-14
  The differences between the perimeter and area of the fovea avascular zone（FAZ） of the carotid artery stenosis side before and after interventional surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ophthalmology and neurology at Qilu Hospital of Shandong University, Jinan, Shandong, China